CLINICAL TRIAL: NCT05198375
Title: Lung UltrasouNd Guided Surfactant Therapy in Preterm Infants: an International Multicentric Randomized Control Trial (LUNG Study)
Brief Title: Lung UltrasouNd Guided Surfactant Therapy in Preterm Infants (LUNG Study)
Acronym: LUNG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility (based on interim analysis)
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Iuri Corsini, Neonatologist at the Careggi University Hospital NICU, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302/2021
Record Dates: First submitted 2021-12-25; First posted 2022-01-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (CG) (Active Comparator): decision to administer exogenous surfactant when FiO2 >0.30 on nCPAP (pressure 6-8 cmH20) to maintain preductal SpO2 between 90 and 95%.
  Interventions: Diagnostic Test: Lung ultrasound score (LUS)
- LUS group (LUSG) (Experimental): decision to administer surfactant when LUS > 8 on nCPAP (pressure 6-8 cmH20) to maintain preductal SpO2 between 90 and 95%.
  The LUS group will receive surfactant administration as rescue therapy in case of LUS < or = 8 but FiO2 > 0.30 on nCPAP (pressure 6-8 cmH20) to maintain preductal SpO2 between 90 and 95%.
  Interventions: Diagnostic Test: Lung ultrasound score (LUS)

INTERVENTIONS:
Diagnostic Test: Lung ultrasound score (LUS) — LU score (LUS) will be performed between 1 and 3 hours of life. LUS will be calculated by performing longitudinal scans of the chest in the anterior (midclavicular line), lateral (anterior axillary line) and posterior (posterior axillary line) area bilaterally using high-frequency linear or micro linear (hockey stick) probe. A score from 0 to 3 will be assigned to each area based on the ultrasound detected pattern.

SUMMARY:
The investigators hypothesized that the use of lung ultrasound (LU) for measuring RDS severity and deciding surfactant treatment thresholds might decrease the incidence of early and late sequelae in the study group. Thus, a timely surfactant therapy would eventually improve short (e.g. Need of mechanical ventilation in the first 3 days) and more long-term outcomes, such as BPD or death.

To confirm this hypothesis, the investigators planned an international multicenter randomized controlled study in which preterm infants will be randomized into two groups: one will be managed deciding surfactant treatment of preterm infants with RDS on the basis of a cut-off value of FiO2 as for European guidelines, and one will be managed deciding surfactant treatment using a LU score cut-off and/or FiO2.

Primary endpoint will be the reduction in proportion of infants with BPD or death in the group managed with LU compared to the control group

DETAILED DESCRIPTION:
Background Management of neonatal respiratory distress syndrome (RDS) involves noninvasive respiratory supports, such as nasal continuous positive airway (nCPAP), and mechanical ventilation. On the other hand, exogenous surfactant administration is the other cornerstone for the treatment of RDS. Currently, the decision to administer surfactant in a non-invasively ventilated newborn is commonly based on cut-off values of inspired fraction of oxygen (FiO2). Nevertheless, the accuracy of this criterion might be weak because FiO2 values depend per se by the setting of respiratory support. Moreover, the American Academy of Pediatrics guidelines do not recommend any FiO2 threshold for surfactant administration. It has been shown that prompt administration of surfactant (within the first 3 hours of life) can reduce the risk of bronchopulmonary dysplasia (BPD). Unfortunately, criteria for surfactant treatment used, often leads to a delayed administration. The role of lung ultrasound (LU) as a semi-quantitative method for the decision to give exogenous surfactant has been studied in recent years. Researchers demonstrated that a LU score (LUS) of RDS severity is able to predict the need for surfactant therapy, as subsequently confirmed by subsequent studies. After these results, a first quality improvement study demonstrated that the use of a LUS cut-off for deciding surfactant treatment allowed a significant increase of early administration. This finding has been confirmed by a recent single-center randomized controlled trial. However, all these studies were single-center, and there are not multicenter randomized controlled trials which can support the wide use of LUS measurement as a standard method for surfactant replacement therapy.

This study, in addition to investigating the decision-making role of LUS in the administration of surfactant, also aims to evaluate the possibility of making treatment with surfactant earlier and more timely, having already been shown in the past that an early administration improves clinical outcomes.

Aim of the study The investigators hypothesized that the use of a LUS for measuring RDS severity and deciding surfactant treatment thresholds might decrease the incidence of early and late sequelae in the study group. Thus, a timely surfactant therapy would eventually improve short (e.g. Need of mechanical ventilation in the first 3 days) and more long-term outcomes, such as BPD or death.

To confirm this hypothesis, the investigators planned an international multicenter randomized controlled study in which preterm infants will be randomized into two groups: one will be managed deciding surfactant treatment of preterm infants with RDS on the basis of a cut-off value of FiO2 (CG), and one will be managed deciding surfactant treatment using a LUS cut-off and FiO2 (LUSG).

Study design The study will be a multicenter randomized open control trial carried out in Level III-IV neonatal intensive care units (NICUs). The financial outcome of the study is no profit. The design of the study is of superiority. The enrollment period will be 24 months (starting February 1, 2022).

Study population The study will take place within the NICUs and therefore in a hospital setting. The study will be multicenter.

The total number of enrolled infants will be 668 (334 per arm). Each center will have to enroll a minimum of 10 children and a maximum of 70.

An interim analysis will be conducted after 167 infants enrolled in each arm (334 total infants enrolled).

Management in the delivery room and in the first hour of life Positive pressure with a neonatal mask and a T-piece system (Neopuff Infant Resuscitator ®, Fisher and Paykel, Auckland, New Zealand) will be used to stabilize the newborns after birth as per routine daily practice. If necessary, infants will start mechanical ventilation in agreement with the European guidelines on neonatal resuscitation. In this latter case the babies will be excluded from the study (see Exclusion criteria section).

In order to better standardize the timing of care after birth, it is expected that assistance in the delivery room, transfer of the newborn to the intensive care unit, stabilization of the newborn and the related procedures (positioning of the vascular access, stabilization of ventilatory parameters, thermal stabilization, etc.) are completed within the first hour of life.

Once infants with RDS have been screened, enrolled in the study, and allocated to the CG or LUSG, LU will be performed as soon as possible between 1 and 3 hours life (<3 h of life). In the meantime, the newborns will be assisted in noninvasive ventilation (nCPAP, pressure 6-8 cmH20) and oxygen to maintain preductal oxygen saturation (SpO2) between 90 and 95%. A loading dose of caffeine citrate of 20 mg/kg will be administered in the first hours of life followed by a maintenance of 5 mg/kg/day, as per routine clinical practice.

Noninvasive ventilation management after the first 3 hours of life or after surfactant administration After the first three hours of life or after having administered surfactant, according to the criteria provided by the randomization group, the newborns can be assisted with non-invasive ventilation other than nCPAP (NIPPV, BiPAP, HFNC) according to the care protocol of the centers involved in the study.

Lung ultrasound procedure LU will be performed by the attending physician. Centers participating to the study should be routinely using LU and all the physician are already trained for the use of the technique.

LUS will be calculated by performing longitudinal scans of the chest in the anterior (midclavicular line), lateral (anterior axillary line) and posterior (posterior axillary line) area bilaterally using high-frequency linear or micro linear (hockey stick) probe between 1 and 3 hour of life. The focus will be located at the level of the pleural line. A score from 0 to 3 will be assigned to each scan area based on the ultrasound detected pattern (in case of different score pattern in the same area the worst will be the one chosen).

LU can be performed keeping the patient in the supine position without the need to rotate him as the posterior axillary line is accessible from the side of the newborn.

Surfactant replacement therapy should be given if LUS is 9 or more in the babies recruited to the LUSG.

The LUS group will receive as rescue therapy surfactant administration in case of LUS < or = 8 but FiO2> 0.30 on nCPAP (pressure 6-8 cmH20) to maintain preductal SpO2 between 90 and 95%.

Surfactant treatment Once criteria for surfactant administration have been reached, surfactant (Curosurf ®, Chiesi, Parma, Italy) will be given (200 mg/kg) according to the InSURE (Intubate-SURfactant-Extubate), LISA (Less- Invasive-Surfactant-Administration) or IN-REC-SURE (INtubate-RECruit-SURfactant-Extubate) technique in both the groups as per the enrollment center protocol.

Pharmacological premedication with fentanest and/or atropine will be allowed (as per center protocol) and recorded.

After surfactant administration, the babies of both groups will be extubated if it has been performed the InSURE or IN-REC-SURE method within 30 min (if satisfactory respiratory drive is present) and will receive nCPAP (pressure 6-8 cmH2O) as per center protocol .

Infants of both groups can receive a subsequent dose of surfactant (100 mg/kg of poractant alfa) using the same method if they meet the non-invasive ventilation failure criteria again during the following 12 to 24 h.

nCPAP ventilation failure criteria In the NICU, nCPAP will be the standard method of noninvasive support in all infants recruited to this trial. nCPAP failure is defined if any of the following criteria are met: FiO2 ≥ 0.30 to maintain a SpO2> 90 for at least 30 min unless rapid clinical deterioration has occurred; respiratory acidosis defined as pCO2 > 65 mmHg (8.5 kPa) and pH <7.20 on an arterial or capillary blood gas sample; apnea defined as more than four episodes of apnea per hour or more than two episodes of apnea per hour when ventilation with bag and mask or Neopuff will be required.

Mechanical ventilation should commence if the patient meets one of the following criteria after additional dose of surfactant: pCO2 > 65 mmHg and pH <7.20, or paO2 <50 mm Hg, or FiO2 >0.40 after surfactant administration or in case of apnea (> 4 episodes in 1 hour or > 2 episodes in 1 hour ventilation with bag and mask or Neopuff ), and should continue with the aim of maintaining a pCO2 of 55-65 mmHg and a SpO2 of 90-95%, using synchronized Mechanical Ventilation (MV), volume controlled MV, or high frequency ventilation.

Patients will be extubated as per center protocol.

ELIGIBILITY:
Inclusion Criteria:

1. In-born infants at 25+0-29+6 weeks of gestational age
2. Spontaneously breathing at birth but requiring noninvasive respiratory support with nCPAP at a pressure of 6-8 cmH2O to maintain an SpO2 between 90% and 95%.
3. Parental consent has been obtained
4. Exclusion of causes of respiratory failure other than RDS

Exclusion Criteria:

1. Endotracheal intubation in the delivery room for resuscitation or insufficient respiratory drive according to European guidelines
2. Prolonged premature rupture of membranes (PROM) for more than 3 days
3. Presence of major congenital malformations or chromosomal anomalies
4. Hydrops fetalis
5. Inherited disorders of metabolism
6. Administration of surfactant before performing the LUS.
7. Other respiratory diseases than RDS

Ages: 1 Minute to 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 411 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
BPD or Death reduction | 36 weeks of gestational age or at the moment of discharge
  Primary endpoint will be the difference in proportion of infants with BPD (defined as Bancalari, Jobe 2001) or death in the group managed with LUS compared to the control group.

SECONDARY OUTCOMES:
Proportion of infants treated "early" (before 3 hours of life) vs late | First 3 hours of life
  Percent of infants treated within 3 hours of life vs late
Age in minute at the first surfactant administration | First 12 hours of life
  Minutes
Needs of mechanical ventilation in the first 3 days of life | First 3 days of life
  Percent of infants needed mechanical ventilation within 3 days of life
Max FiO2 value before surfactant treatment | First 12 hours of life
  FiO2 value
FiO2/SpO2 ratio before surfactant treatment | First 12 hours of life
  FiO2/SpO2 ratio
Duration of non-invasive and invasive respiratory support (included O2 therapy) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Days
Proportion of infants needed to receive multiple doses of surfactant | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Duration of hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Days
Occurrence of BPD using multiple definitions | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Proportion
Proportion of infants with patent ductus arteriosus treated pharmacologically and/or surgically | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Proportion of infants with pneumothorax | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Proportion of infants with retinopathy of prematurity | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Proportion of infants with intraventricular hemorrhage > or = grade 3 | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Proportion of infants with periventricular leukomalacia | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Proportion of infants with necrotizing enterocolitis > stage 2 | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Use of systemic postnatal steroids | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Mortality | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage
Pulmonary hemorrhage | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Iuri Corsini, MD, Principal Investigator — Careggi University Hospital of Florence
Locations (18):
- Italy (12):
  - Neonatal intensive care unit - Azienda Sanitaria dell'Alto Adige, Bolzano
  - Spedali Civili di Brescia, Brescia
  - AOU Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano, Milan
  - Neonatal Intensive Care Unit Ospedale dei Bambini "Vittore Buzzi", Milan
  - Neonatal Intensive Care Unit Modena, Modena
  - Neonatal Intensive Care Unit - Federico II University, Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Neonatologia e Terapia Intensiva Neonatale Rimini, Rimini
  - Fondazione Policlinico Gemelli, Roma
  - Azienda sanitaria universitaria Friuli Centrale, Udine
  - NICU AOUI Verona, Verona
- Spain (6):
  - Germans Trias i Pujol, Badalona, Spain
  - Neonatal Intensive Care Unit Coruña, A Coruña
  - Barcelona Center for Maternal Fetal and Neonatal Medicine, Barcelona
  - Neonatal Intensive Care Unit, Puerta del Mar Universitary Hospital, Cádiz., Cadiz
  - Hospital Gregorio Maranon, Madrid
  - Hospital Alvaro Cunqueiro de Vigo. Instituto de Investigación Galicia Sur, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Bahadue FL, Soll R. Early versus delayed selective surfactant treatment for neonatal respiratory distress syndrome. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD001456. doi: 10.1002/14651858.CD001456.pub2. PMID 23152207
- [Background] Raschetti R, Yousef N, Vigo G, Marseglia G, Centorrino R, Ben-Ammar R, Shankar-Aguilera S, De Luca D. Echography-Guided Surfactant Therapy to Improve Timeliness of Surfactant Replacement: A Quality Improvement Project. J Pediatr. 2019 Sep;212:137-143.e1. doi: 10.1016/j.jpeds.2019.04.020. Epub 2019 May 10. PMID 31079857
- [Background] Rodriguez-Fanjul J, Jordan I, Balaguer M, Batista-Munoz A, Ramon M, Bobillo-Perez S. Early surfactant replacement guided by lung ultrasound in preterm newborns with RDS: the ULTRASURF randomised controlled trial. Eur J Pediatr. 2020 Dec;179(12):1913-1920. doi: 10.1007/s00431-020-03744-y. Epub 2020 Jul 24. PMID 32710304
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Background] De Martino L, Yousef N, Ben-Ammar R, Raimondi F, Shankar-Aguilera S, De Luca D. Lung Ultrasound Score Predicts Surfactant Need in Extremely Preterm Neonates. Pediatrics. 2018 Sep;142(3):e20180463. doi: 10.1542/peds.2018-0463. Epub 2018 Aug 14. PMID 30108142
- [Background] De Luca D, van Kaam AH, Tingay DG, Courtney SE, Danhaive O, Carnielli VP, Zimmermann LJ, Kneyber MCJ, Tissieres P, Brierley J, Conti G, Pillow JJ, Rimensberger PC. The Montreux definition of neonatal ARDS: biological and clinical background behind the description of a new entity. Lancet Respir Med. 2017 Aug;5(8):657-666. doi: 10.1016/S2213-2600(17)30214-X. Epub 2017 Jul 4. PMID 28687343
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Corsini I, Parri N, Ficial B, Dani C. Lung ultrasound in the neonatal intensive care unit: Review of the literature and future perspectives. Pediatr Pulmonol. 2020 Jul;55(7):1550-1562. doi: 10.1002/ppul.24792. Epub 2020 Apr 27. PMID 32339409
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Raimondi F, Migliaro F, Corsini I, Meneghin F, Pierri L, Salome S, Perri A, Aversa S, Nobile S, Lama S, Varano S, Savoia M, Gatto S, Leonardi V, Capasso L, Carnielli VP, Mosca F, Dani C, Vento G, Dolce P, Lista G. Neonatal Lung Ultrasound and Surfactant Administration: A Pragmatic, Multicenter Study. Chest. 2021 Dec;160(6):2178-2186. doi: 10.1016/j.chest.2021.06.076. Epub 2021 Jul 19. PMID 34293317
- [Background] Raimondi F, Migliaro F, Corsini I, Meneghin F, Dolce P, Pierri L, Perri A, Aversa S, Nobile S, Lama S, Varano S, Savoia M, Gatto S, Leonardi V, Capasso L, Carnielli VP, Mosca F, Dani C, Vento G, Lista G. Lung Ultrasound Score Progress in Neonatal Respiratory Distress Syndrome. Pediatrics. 2021 Apr;147(4):e2020030528. doi: 10.1542/peds.2020-030528. Epub 2021 Mar 9. PMID 33688032
- [Background] de Vries LS, Eken P, Dubowitz LM. The spectrum of leukomalacia using cranial ultrasound. Behav Brain Res. 1992 Jul 31;49(1):1-6. doi: 10.1016/s0166-4328(05)80189-5. PMID 1388792
- [Background] International Committee for the Classification of Retinopathy of Prematurity. The International Classification of Retinopathy of Prematurity revisited. Arch Ophthalmol. 2005 Jul;123(7):991-9. doi: 10.1001/archopht.123.7.991. PMID 16009843
- [Background] Bell MJ, Ternberg JL, Feigin RD, Keating JP, Marshall R, Barton L, Brotherton T. Neonatal necrotizing enterocolitis. Therapeutic decisions based upon clinical staging. Ann Surg. 1978 Jan;187(1):1-7. doi: 10.1097/00000658-197801000-00001. PMID 413500
- [Derived] Corsini I, Rodriguez-Fanjul J, Raimondi F, Boni L, Berardi A, Aldecoa-Bilbao V, Alonso-Ojembarrena A, Ancora G, Aversa S, Beghini R, Meseguer NB, Capasso L, Chesi F, Ciarcia M, Concheiro A, Corvaglia L, Ficial B, Filippi L, Carballal JF, Fusco M, Gatto S, Ginovart G, Gregorio-Hernandez R, Lista G, Sanchez-Luna M, Martini S, Massenzi L, Miselli F, Mercadante D, Mosca F, Palacio MT, Perri A, Piano F, Prieto MP, Fernandez LR, Risso FM, Savoia M, Staffler A, Vento G, Dani C. Lung UltrasouNd Guided surfactant therapy in preterm infants: an international multicenter randomized control trial (LUNG study). Trials. 2023 Nov 4;24(1):706. doi: 10.1186/s13063-023-07745-8. PMID 37925512